CLINICAL TRIAL: NCT02300961
Title: A Risk Stratification Model for Neurocognitive Outcome After Transplant and Feasibility of an Early Cognitive Intervention Program
Brief Title: Feasibility Neurocognitive Outcome After Transplant
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-31680; NCI-2014-02434 (Other: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stem Cell Transplantation; Pediatric Cancer; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive rehabilitation arm (Experimental): Cognitive rehabilitation program
  Interventions: Behavioral: Cognitive rehabilitation program

INTERVENTIONS:
Behavioral: Cognitive rehabilitation program

SUMMARY:
This pilot study will primarily be evaluated by feasibility and adherence to an iPad-based neurocognitive intervention program. It will secondarily be evaluated by performance on the neurocognitive testing post-transplant and change in performance in subsequent years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a histologic or cytological diagnosis of ALL treated with stem cell transplantation. There are no restrictions on prior therapy.
* Patients must be between the ages of 6 years and 21 years of age (inclusive), but there will be no discrimination based on gender, race, creed, or ethnic background. The age limits are set at 6 years of age in order to ensure that patients will be able to participate in these specific cognitive rehabilitation tasks. ECOG/KPS will not be employed.
* Patient and/or parents/guardians as appropriate must sign an informed consent, be mentally responsible, able to understand and willing to sign a written informed consent.

Exclusion Criteria:

* Subjects with significant concurrent medical complications that in the judgment of the Principal Investigator(s) could affect the patient's ability to complete the planned trial. There are no therapy restrictions or restrictions regarding the use of other Investigational Agents.
* Pregnant patients will be excluded.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete the post-transplant neurocognitive intervention program | 3 months after enrollment
  Number of participants who enroll in and are able to complete the neurocognitive intervention program, measured at 3 months after enrollment.

SECONDARY OUTCOMES:
Number of participants who complete at least half of the neurocognitive intervention program | 3 months after enrollment
  Number of participants who complete at least 50% of scheduled sessions in the neurocognitive intervention program.
Change in WISC-IV or WAIS-IV scores | Baseline, 1 year post-treatment, 2 years post-treatment
  Change in intellectual functioning scores (Full Scale IQ, Verbal Comprehension, Perceptual Reasoning, Working Memory, and Processing Speed indices) from pre-treatment to 1 and 2 years post-treatment.
Change in WRAML-2 scores | Baseline, 1 year post-treatment, 2 years post-treatment
  Change in verbal and visual memory scores from pre-treatment to 1 and 2 years post-treatment using the Wide Range Assessment of Memory and Learning, Second Edition (WRAML-2).
Change in executive functioning scores (D-KEFS or NEPSY-II) | Baseline, 1 year post-treatment, 2 years post-treatment
  Change in executive functioning scores from pre-treatment to 1 and 2 years post-treatment, using Delis Kaplan Executive Function System (D-KEFS; ages 8-21) or NEPSY-II subtests (ages 6-7).
Change in CPT-II scores | Baseline, 1 year post-treatment, 2 years post-treatment
  Change in sustained attention/vigilance scores from pre-treatment to 1 and 2 years post-treatment using Conners' Continuous Performance Test, Second Edition (CPT-II).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hiniker, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No